CLINICAL TRIAL: NCT05034224
Title: MACCUS: ModulAtion of Cardiac Coronary Sinus Hemodynamics to Develop a New Treatment for microvascUlar diseaSe. A Single Center, Randomized Study.
Brief Title: Coronary Sinus Pressure and Microvascular Disease
Acronym: MACCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Clinical Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021-4
Record Dates: First submitted 2021-08-23; First posted 2021-09-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Microvascular Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The study is a single-center, cross-over randomized trial to investigate the effect of coronary sinus occlusion on microvascular resistances.
Who Masked: Participant, Investigator
Masking Description: Investigators performing the analysis of the data (post-hoc) and patients are blinded to the sequence of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): The index of microvascular resistances will be measured while a balloon placed in the coronary sinus is kept deflated.
  Interventions: Device: Swan-Ganz catheter placed in the coronary sinus - deflated
- Coronary sinus occlusion (Active Comparator): The index of microvascular resistances will be measured while a balloon placed in the coronary sinus is inflated.
  Interventions: Device: Swan-Ganz catheter placed in the coronary sinus - inflated

INTERVENTIONS:
Device: Swan-Ganz catheter placed in the coronary sinus - deflated — A normal Swan-Ganz catheter will be advanced in the coronary sinus. The Balloon will be kept deflated during sham intervention. The index of microvascular resistances will be measured using the Abbott Pressure Wire X as per instructions for use durng both interventions.
  Arms: Sham
Device: Swan-Ganz catheter placed in the coronary sinus - inflated — A normal Swan-Ganz catheter will be advanced in the coronary sinus. The Balloon will be inflated to obtain coronary sinus occlusion during the active intervention. The index of microvascular resistances will be measured using the Abbott Pressure Wire X as per instructions for use durng both interventions.
  Arms: Coronary sinus occlusion

SUMMARY:
MACCHUS is a randomized, single-center, controlled, cross-over interventional study in which coronary artery resistances will be measured at baseline and during temporary occlusion of the coronary sinus.

DETAILED DESCRIPTION:
The aim of this study is to test whether an increase in coronary sinus pressure leads to a change in coronary microvascular resistances in patients with angina pectoris and with an indication to measurement of microvascular function as per clinical guidelines.

All patients with a clinical indication for the assessment of microvascular function will be invited to participate and will sign the informed consent at least 24 hours before the study. Patients with an index of microvascular resistances >25 (i.e. evidence of microvascular dysfunction) will undergo study-specific procedures in the same session (i.e. no additional invasive procedure is required for the study).

Study-specific procedures include the repetition of the assessment of microvascular resistances at rest and during coronary sinus occlusion. Coronary sinus occlusion will be achieved by inflating a balloon sized to ~70% of the diameter of the coronary sinus. Since the implantation of a coronary sinus reducer is a therapeutic option for this type of patients, also this procedure (inflation of an undersized balloon in the coronary sinus) provides clinically relevant information (sizing of the vessel, effect on microvascular resistances and feasibility of the intervention).

The primary goal of the study is to study the effect of coronary sinus occlusion on microvascular resistances at rest and during hyperemia.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome (including patients with anginal equivalents).
* Reversible ischemia on non-invasive testing, indication to cardiac catheterization;
* Indication to the assessment of microvascular function (note: patients will be asked for participation and consented prior to the first measurement of microvascular function, which will be conducted as per clinical indication; only those with evidence of pure or mixed microvascular disease (index of microvascular resistances (IMR)>25 will proceed into the study);
* Willingness to participate and ability to understand, read and sign the informed consent;
* Age>18 years

Exclusion Criteria:

* Previous CABG with patent grafts to the left anterior descending coronary
* Epicardial coronary disease (FFR <0.80 with evidence of a focal stenosis) in the left anterior descending territory
* Severe valvular heart disease
* Any cardiomyopathy; pulmonary or renal disease
* Inability to provide informed consent
* Any disease reducing life expectancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Index of microvascular resistances (balloon occlusion versus deflated balloon) | 1 Minute after balloon occlusion
  The Index of microvascular resistances, calculated as (Pressure distal - coronary venous pressure ) x mean transit time, will be compared between the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ullrich H, Hammer P, Olschewski M, Munzel T, Escaned J, Gori T. Coronary Venous Pressure and Microvascular Hemodynamics in Patients With Microvascular Angina: A Randomized Clinical Trial. JAMA Cardiol. 2023 Oct 1;8(10):979-983. doi: 10.1001/jamacardio.2023.2566. PMID 37610757
- [Derived] Ullrich H, Olschewski M, Munzel T, Gori T. Randomized, crossover, controlled trial on the modulation of cardiac coronary sinus hemodynamics to develop a new treatment for microvascular disease: Protocol of the MACCUS trial. Front Cardiovasc Med. 2023 Feb 16;10:1133014. doi: 10.3389/fcvm.2023.1133014. eCollection 2023. PMID 36873411